CLINICAL TRIAL: NCT06808555
Title: Pai.ACT: An Artificial Intelligence-Driven Chatbot-Assisted ACT Mobile Platform With Mental Health Triage - A Randomized Controlled Trial and Regional Service Evaluation
Brief Title: Pai.ACT: AI-Driven ACT Chatbot for Mental Health Triage and Service Evaluation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Social Welfare Department, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20250114-002-000
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Disorder With Hyperactivity (ADHD); Neurodevelopmental Disorder (Diagnosis); Dyslexia
Keywords: Smartphone-delivered Therapy; Deep learning; Acceptance and Commitment Therapy; Parents; Children with Special Needs; Parental Support; Artificial Intelligence in Healthcare; Psychological Interventions; Parenting Stress; Regional Randomized Controlled Trial
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders; Disease; Dyslexia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to either the Pai.ACT Group or Control Group in a 1:1 ratio using a permuted block size of 6, stratified by child's age (preschool, school age). Randomization will utilize sequentially numbered, opaque, sealed envelopes with number cards (1=intervention, 2=control), prepared by clerical staff uninvolved in the study. An independent statistician will generate and conceal randomization details from the research team. Following informed consent and baseline assessments, a blinded research assistant will open the envelopes. Both groups will access their respective interventions through a secure e-link, using unique login credentials tied to their mobile device's ID, accompanied by weekly reminders. The Pai.ACT application includes content-locking features to prevent sharing of its audio and video materials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pai.ACT Group (Experimental): Parents allocated to this experimental group will gain complete access to the Pai.ACT mobile app.
  Interventions: Behavioral: Pai.ACT Group
- Control Group (Other): Parents allocated to the Control Group will receive standard family support through Hong Kong's family and children rehabilitation services, which are administered by government-funded units under the Social Welfare Department. Parents will participate in structured psychoeducation sessions focusing on positive parenting and will have access to peer support groups, while their children will receive individualized training plans tailored for neurodevelopmental conditions, in addition to referrals for speech and occupational therapy.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Pai.ACT Group — The Pai.ACT mobile app is an innovative therapeutic tool that utilizes Acceptance and Commitment Therapy (ACT). It integrates a sophisticated AI algorithm to analyze self-reported data and conversation texts when the user interacts with the AI chatbot and identifies what psychological inflexibility processes are required to be the most essential to be addressed for process-matched ACT interventions. Following interactions with the AI chatbot, Pai.ACT provides a stratified mental health support, categorizing into three risk levels:
  * Low-risk: Users access self-help ACT digital modules tailored to their specific psychological inflexibility processes.
  * Moderate-risk: In addition to the self-help modules, users receive 4-6 sessions of video-conferencing-based ACT interventions (45-60 minutes per session) conducted by our trained counseling team.
  * High-risk: Users are directed to specialized mental health services provided by collaborating units.
  Arms: Pai.ACT Group
Other: Control Group — Both the Pai.ACT intervention group and the control group will receive standard family support through Hong Kong's family and children rehabilitation services, which are administered by government-funded units under the Social Welfare Department. Parents will participate in structured psychoeducation sessions focusing on positive parenting and will have access to peer support groups. Their children will receive individualized training plans tailored for neurodevelopmental conditions, in addition to referrals for speech and occupational therapy.
  Arms: Control Group

SUMMARY:
Parents of children with special needs in Hong Kong often face limited psychological support, which can negatively impact the child rehabilitation process and the well-being of parent-child relationships. To address this gap, we have developed Pai.ACT, the first deep learning-based mental health advisory system for parents.

Pai.ACT features an AI chatbot that integrates the counselling principles of Acceptance and Commitment Therapy (ACT) through natural language processing, providing parents with a human-like voice-to-text experience. Using data from chatbot interactions, the Pai.ACT platform offers assessments regarding the individual's psychological inflexibility status and delivers stratified mental health interventions by:

* Low-risk: Users access self-help ACT digital modules tailored to their specific psychological inflexibility processes.
* Moderate-risk: In addition to the self-help modules, users receive 4-6 sessions of video-conferencing-based ACT interventions (45-60 minutes per session) conducted by our trained counseling team.
* High-risk: Users are directed to specialized mental health services provided by collaborating units.

The study includes a regional randomised controlled trial (RCT) in Hong Kong's Sha Tin District, in collaboration with the Shatin District Office. The goal of this regional study is to evaluate the feasibility, acceptability, and potential efficacy of combining AI-driven mental health support across all of Hong Kong. Focus group interviews will also explore parents' perceptions of Pai.ACT and help identify the most effective service model for scaling its use.

Pai.ACT provides accessible and comprehensive mental health services to Chinese-speaking parents, helping to alleviate the psychological burden of caregiving. By integrating mental health support with child rehabilitation services and non-governmental organisations, Pai.ACT has the potential to enhance family caregivers' well-being, reduce stigma associated with special needs children, and promote more significant mental health awareness in Chinese-speaking communities.

DETAILED DESCRIPTION:
Introduction Children with special needs include those with chronic developmental, behavioural, or emotional conditions requiring specialised and prolonged health services beyond those typically required by children. In Hong Kong, common conditions include autism spectrum disorders (ASD), attention-deficit hyperactivity disorder (ADHD), and developmental disabilities or delays. Over recent years, the prevalence of children with special needs has risen significantly. In 2019, the Child Assessment Centre under the Department of Health reported annual increases of 6.2% to 10.7% in newly diagnosed cases and referrals for specialised follow-up services for preschool-aged children.

Despite the growing demand, Hong Kong's existing health and social services for children with special needs face several challenges. Prolonged waiting times for multidisciplinary assessments, diagnoses, and intensive rehabilitation services delay critical support and exacerbate the psychological burden on parents. Without a certified diagnosis from mental health professionals, parents often struggle to access public health services for rehabilitation, leaving them unsupported during crucial stages of caregiving.

The local mental health system primarily focuses on severe mental illnesses, with limited resources dedicated to the psychological well-being of parents. Parents of children with special needs face additional barriers to accessing mental health services, including time constraints, caregiving responsibilities, geographic limitations, and a scarcity of professionals trained to address their unique challenges. Furthermore, self-stigma often prevents parents from seeking help, even when they recognise the impact of poor mental health on their caregiving abilities. As a result, parents of children with special needs report higher levels of parenting stress and depressive symptoms compared to parents of neurotypical children.

Acceptance and Commitment Therapy (ACT) Acceptance and Commitment Therapy (ACT) has emerged as an effective psychotherapy for addressing parenting challenges. ACT helps individuals develop cognitive defusion, acceptance, and value clarification skills, allowing them to manage distressing emotions better and reconnect with their caregiving values. Research has shown that ACT significantly improves psychological well-being and reduces somatic complaints in diverse populations. Recent clinical trials targeting paediatric conditions such as ASD, asthma, cerebral palsy, and acquired brain injury have demonstrated significant reductions in parenting stress, depression, and anxiety symptoms.

Despite its effectiveness, traditional in-person delivery of ACT poses challenges for parents of children with special needs due to time constraints and caregiving responsibilities. The COVID-19 pandemic has further highlighted the need for virtual healthcare options, with smartphone-based ACT platforms emerging as a viable solution. Smartphone-based interventions offer parents convenient access to ACT, overcoming geographical and time-related barriers while reducing the resource demands on healthcare systems. Studies have shown that parents are open to incorporating technology into their care, with smartphone-based ACT interventions demonstrating improvements in psychological flexibility, well-being, mindfulness skills, and children's quality of life.However, maintaining long-term engagement with mental health apps remains a challenge. Studies indicate that over 70% of users discontinue use shortly after downloading such applications. This highlights the need for innovative and engaging approaches to sustain user participation and maximise the impact of digital mental health interventions.

Pai.ACT

Pai.ACT is an innovative smartphone application designed to enhance the well-being of parents with children who have special needs. The application merges artificial intelligence (AI) technology with Acceptance and Commitment Therapy (ACT) principles to offer personalized psychological support. The core feature of Pai.ACT is an AI-driven chatbot with voice-to-text capabilities, which delivers responses from ACT counselors in Cantonese, thus enabling human-like interactions. This chatbot is powered by a patented AI model that has been trained on over 19,000 annotated ACT session texts to ensure accurate and contextually relevant psychotherapeutic interactions, as well as to assess a user's psychological inflexibility through real-time textual analysis. Following interactions with the AI chatbot, Pai.ACT provides a tiered mental health support system tailored to the specific needs of parents, categorized into three risk levels:

* Low-risk: Users access self-help ACT digital modules tailored to their specific psychological inflexibility processes.
* Moderate-risk: In addition to the self-help modules, users receive 4-6 sessions of video-conferencing-based ACT interventions (45-60 minutes per session) conducted by our trained counseling team.
* High-risk: Users are directed to specialized mental health services provided by collaborating units.

This comprehensive, multi-tiered approach optimizes resources and ensures timely and effective mental health support for parents.

Study aim and hypotheses This study evaluates the feasibility, acceptability, and preliminary efficacy of Pai.ACT, a scalable digital mental health intervention designed for parents of children with special needs in Hong Kong. A randomized controlled trial (RCT), conducted in collaboration with the Sha Tin District Office, will assess the intervention's potential for citywide implementation. The regionally delimited trial (Sha Tin District) will serve as a proof-of-concept, with outcomes informing adaptations for broader dissemination across Hong Kong's diverse administrative regions. It is hypothesized that, compared to the control group receiving standard parenting advice, parents who engage with Pai.ACT will experience significant improvements in mental well-being and psychological flexibility, alongside reductions in the emotional and behavioral symptoms of their children with special needs.

Significance of the Study If successful, Pai.ACT could serve as a scalable and effective mental health solution for parents of children with special needs, addressing a critical gap in Hong Kong's healthcare system. By leveraging AI-driven technology, the platform offers an accessible, cost-effective, and flexible intervention that aligns with the caregiving demands of parents. Beyond improving parental mental health, the integration of Pai.ACT with existing child rehabilitation services could lead to broader societal benefits, including reduced stigma associated with special needs children and increased mental health awareness in Hong Kong.

This study will provide key insights into the feasibility of combining AI-driven mental health interventions with existing healthcare systems, paving the way for future large-scale implementations across Hong Kong and beyond.

ELIGIBILITY:
Inclusion Criteria:

The participants of the study are primary caregivers, specifically parents, must be Cantonese-speaking residents of Hong Kong.

Eligible parents are required to cohabitate with a child aged 2 to 9 years who has either a confirmed or suspected diagnosis of a neurodevelopmental condition, including Autism Spectrum Disorder (ASD), Attention-Deficit/Hyperactivity Disorder (ADHD), or Developmental Delay (DD). These conditions must be recognised by the Child Assessment Service of the Department of Health and meet the diagnostic criteria specified in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). The diagnosis or suspected diagnosis must be formally documented in the child's case profile maintained at the collaborating non-governmental organisations.

Exclusion Criteria:

* Parents diagnosed with severe mental illnesses.
* Pregnant parents or those less than six months postpartum.
* Parents with a developmental disability that impairs their ability to understand the program's content.
* Parents with cognitive, language, communication, visual, or hearing impairments that could hinder their comprehension of the intervention content.
* Parents actively participating in other psychosocial, psychoeducational, or parenting interventions.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress | Change from baseline to immediate and 6 months post-intervention
  Parenting stress will be assessed using the Parental Stress Scale (PSS, 18-item, 5-point scale). The PSS evaluates parental satisfaction and strain regarding parenting roles. A higher score represents a higher level of parental stress. The Chinese PSS version, including its parenting stress, will be assessed using the Parental Stress Scale (PSS), which consists of 18 items and uses a 5-point rating system. The PSS is designed to evaluate how parents perceive their roles in terms of satisfaction and strain. A higher score indicates a greater level of parental stress. The Chinese version of the PSS, along with its subscales, has demonstrated strong validity in terms of both convergent and discriminant measures, as well as good internal consistency, with a Cronbach's alpha ranging from .79 to .88 among Chinese parents.
Child's Emotional and Behavioural Symptoms | Change from baseline to immediate and 6 months post-intervention
  The Strengths and Difficulties Questionnaire (SDQ) is designed to evaluate a child's emotional and behavioral symptoms. It employs a 3-point Likert scale to assess the following areas: emotional symptoms, conduct problems, hyperactivity/inattention, peer problems, and prosocial behavior. Each of these subscales consists of five items. The Chinese version of the SDQ has demonstrated adequate test-retest reliability, with an Intraclass Correlation Coefficient ranging from .75 to .86, and has shown good discriminant validity among parents in Hong Kong.

SECONDARY OUTCOMES:
Depressive Symptoms | Change from baseline to immediate and 6 months post-intervention
  Depressive symptoms will be evaluated using the Patient Health Questionnaire (PHQ-9). The PHQ-9 consists of 9 items on a 4-point Likert scale, with a total score of 10 or higher indicating potential depression.
Anxiety Symptoms | Change from baseline to immediate and 6 months post-intervention
  Anxiety symptoms will be evaluated using the Generalized Anxiety Disorder-7 (GAD-7) scale. The GAD-7 is a 7-item, 4-point Likert scale, where a total score of ≥10 indicates a potential anxiety disorder.
Psychological Flexibility | Change from baseline to immediate and 6 months post-intervention
  Psychological flexibility will be assessed using the Psyflex questionnaire and/or the Comprehensive Assessment of Acceptance and Commitment Therapy (CompACT). The Psyflex is a 6-item, 5-point Likert scale designed to measure psychological flexibility, while the CompACT measures the core processes of ACT, including openness to experience, behavioural awareness, and valued action. Each item is rated on a 7-point Likert scale, with higher scores indicating greater psychological flexibility.
Perceived usability of the mobile app | At immediate post-intervention and 6 months post-intervention
  Perceived usability of the mobile app will be measured using the System Usability Scale (SUS). The SUS is a 10-item, 10-point Likert scale. The total SUS score ranges from 0 to 100. A score of at least 80 out of 100 indicates high perceived usability. This score suggests that the mobile app, integrated with the 'Pai.ACT' mental health advisory system, is highly usable for end users. These end users are primarily parents of children with Special Health Care Needs (SHCN).

IPD SHARING:
Plan to Share IPD: No